CLINICAL TRIAL: NCT07147686
Title: The Effects of Continuous Repetition of Motor Skills at a Consistent Speed With Music on Decision-Making and Independent Learning Abilities in Children Aged 8-9 Years: A Pre/Post-Test Quasi-Experimental Study With Control Group
Brief Title: Does the Continuous Repetition of Motor Skills at a Consistent Speed With Music Affect Children's Decision-Making and Learning Abilities?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bekir tokay (Other)
Collaborators: Uşak University (Other)
Responsible Party: Sponsor-Investigator, bekir tokay, Dr., Lecturer, Uşak University
Organization: Uşak University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-140; 2023-140 (Other: Uşak University Ethics Committee)
Record Dates: First submitted 2025-08-18; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Healhty
Keywords: motor skills; Cognitive Development; music; Decision-Making; Independent Learning; Executive Functions

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group, quasi-experimental design with a pre/post-test structure. Participants were assigned by classroom to one of three groups: Control (no music intervention), Slow Tempo Motor Exercise with music (30 BPM), and Fast Tempo Motor Exercise with music (60 BPM). Each group followed the assigned intervention throughout the 14-week study period. Outcome measures included decision-making and independent learning skills, assessed using validated psychometric scales.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Slow Tempo Group (Experimental): Participants perform motor exercises accompanied by music at 30 beats per minute (BPM) for 14 weeks.
  Interventions: Behavioral: Slow tempo basic motor skills exercises with music (30 BPM)
- Arm 2: Fast Tempo Group (Experimental): Participants perform motor exercises accompanied by music at 60 beats per minute (BPM) for 14 weeks.
  Interventions: Behavioral: Fast tempo basic motor skills exercises with music (60 BPM)
- Arm 3: Control Group: (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Slow tempo basic motor skills exercises with music (30 BPM) — Participants performed basic motor skills exercises synchronized with slow-tempo music at 30 beats per minute (BPM). The slow tempo was intended to enhance internal timing, cognitive inhibition, controlled movement coordination, and sustained attention. Each session lasted 10-15 minutes per exercise, using traditional Turkish music (e.g., Erik Dali, Horon, Sari Zeybek) to provide culturally relevant rhythmic patterns.
  Arms: Arm 1: Slow Tempo Group
Behavioral: Fast tempo basic motor skills exercises with music (60 BPM) — Participants performed basic motor skills exercises synchronized with fast-tempo music at 60 BPM. The faster tempo aimed to increase reaction speed, attention demand, processing speed, decision-making, and cognitive flexibility. Each session lasted 10-15 minutes per exercise, using traditional Turkish music with asymmetric rhythms to challenge timing and planning skills.
  Arms: Arm 2: Fast Tempo Group

SUMMARY:
This study examined whether repeating motor skill exercises at a consistent speed with music can improve decision-making and independent learning abilities in children aged 8-9 years. Children participated in either slow tempo, fast tempo, or no-music control exercise sessions. Music was used to help regulate tempo and attention, and exercises were designed to enhance timing, focus, and planning skills. The study measured cognitive outcomes using validated scales for independent learning and decision-making.

DETAILED DESCRIPTION:
This quasi-experimental study with a control group investigated the effects of continuous motor skill exercises accompanied by music on decision-making and independent learning abilities in children aged 8-9 years. A total of 399 children completed the study (186 females, 213 males), divided into Control (124), Slow Tempo Motor Exercise (140), and Fast Tempo Motor Exercise (135) groups.

Music was integrated into exercises to regulate tempo and cognitive load, enhancing attention, processing speed, timing, and executive functions. Slow tempo exercises (30 BPM) focused on internal timing, cognitive inhibition, and controlled movement coordination. Fast tempo exercises (60 BPM) aimed to improve reaction times, attention, decision-making, and planning. Traditional Turkish music genres (Erik Dali, Horon, Sari Zeybek) were selected to support rhythmic coordination and cultural relevance. Each session lasted 10-15 minutes per exercise.

Two psychometric scales were used:

Scale of Independent Learning Skills (SILS): Measures metacognitive, affective, and cognitive skills (18 items, 4-point Likert scale, Cronbach's α = .81).

Decision-Making Skills Assessment Scale (DMSAS): Evaluates dependent, independent, and ability-based decision-making (17 items, 4-point Likert scale, Cronbach's α = .65-.70).

Scales were administered face-to-face in classrooms by trained interviewers. Participants responded simultaneously, and responses were collected for later evaluation. No personal information was included.

The study aimed to analyze how music and exercise tempo affect children's cognitive functions and executive skills, emphasizing rhythmic coordination, attention, and culturally relevant music.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-9 years.
* Enrolled in school and selected by classroom to prevent contamination between intervention and control groups.
* Written informed consent obtained from parents or legal guardians.
* Able to participate in motor exercises and music-accompanied sessions.
* Understanding of the study purpose and procedures by both child and parent/guardian.

Exclusion Criteria:

* Absence or withdrawal during the study period.
* Serious health problems, chronic illnesses, or physical limitations preventing participation in exercises.
* Withdrawal of consent by participant or parent/guardian.
* Cognitive or attentional difficulties that prevent completion of motor and cognitive tasks.

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 399 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Independent Learning Skills (SILS Total Score) | Baseline and Post-Intervention (14 weeks)
  Independent Learning Skills will be assessed using the Scale of Independent Learning Skills (SILS). Total score will be computed per the instrument manual (4-point Likert for 18 items; reverse-scoring not applicable). Analyses will use change from baseline to 14 weeks.
Decision-Making Skills (DMSAS Total Score) | Baseline and Post-Intervention (14 weeks)
  Decision-Making Skills will be assessed using the Decision-Making Skills Assessment Scale (DMSAS; 17 items; includes reverse-coded items). Total score will be computed per the instrument manual. Analyses will use change from baseline to 14 weeks.

SECONDARY OUTCOMES:
SILS Subscale Scores (Metacognitive, Affective, Cognitive) | Baseline and Post-Intervention (14 weeks)
  Subscale scores of the SILS scale, assessing metacognitive, affective, and cognitive components of learning strategies.
DMSAS Subscale Scores (Decision-Making According to Abilities, Consequences, and Planning) | Baseline and Post-Intervention (14 weeks)
  Subscale scores of the DMSAS scale, assessing decision-making according to abilities, consequences, and planning.

CONTACTS AND LOCATIONS:
Overall Officials: Bekir TOKAY, Ph.D., Principal Investigator — Uşak University; Mustafa AKIL, Prof. Dr., Study Chair — Uşak University
Locations (1):
- Faculty of Sport Sciences, Uşak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared due to the young age of participants and privacy concerns. All collected data are confidential and will only be used for the purposes of this study.